CLINICAL TRIAL: NCT05940584
Title: Implementation and Evaluation of a Tele-reha As Well As a Paper-based Aftercare Programme Following Inpatient Rehabilitation: a Three-armed, Observer-blinded, Randomised Controlled Trial
Brief Title: Tele-reha Versus Paper-based Aftercare Programme Following Inpatient Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Neurologisches Rehabiliationszentrum Rosenhügel (Other)
Responsible Party: Principal Investigator, Valentin Ritschl, Postdoctoral Researcher in Outcomes Research, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRZ_Tele_Reha
Record Dates: First submitted 2023-06-16; First posted 2023-07-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To minimise observer bias, the assessors will be blinded and will have no knowledge of the group allocation. The assessors will only be involved at the assessment time points, but at no other stage of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group Tele-reha (1) (Experimental): Tele-reha group
  Interventions: Device: Tele-Reha provided with EvoPads
- Control Group Paper-based exercises (1) (Active Comparator): Paper-based exercises with option to do tele-reha afterwards
  Interventions: Other: Paper-based exercises with option to do tele-reha afterwards
- Control Group Paper-based exercises (2) (Active Comparator): Only paper-based exercises
  Interventions: Other: Only paper-based exercises

INTERVENTIONS:
Device: Tele-Reha provided with EvoPads — Exercises and cognitive training provided on an EvoPad
  Arms: Intervention Group Tele-reha (1)
Other: Paper-based exercises with option to do tele-reha afterwards — Similar exercises and cognitive training as Group 1 provided on paper. Patients receive the Tele-Reha afterwards
  Arms: Control Group Paper-based exercises (1)
Other: Only paper-based exercises — Same exercises and cognitive training as Group 2 provided on paper only.
  Arms: Control Group Paper-based exercises (2)

SUMMARY:
The goal of this three-armed, observer-blinded, randomised controlled trial is to (i) to implement a telerehabilitation intervention in routine care after an inpatient rehabilitation stay for people insured with the Social Insurance Institution for the Self-Employed (SVS), (ii) to evaluate the impact of telerehabilitation on the consolidation of goals achieved during the inpatient stay in everyday life, and (iii) to evaluate whether independence in everyday life can be increased by implementing telerehabilitation at home compared to standard care. Our hypothesis is that the tele-reha intervention, including ongoing therapist support, will improve independence in daily living (defined as the primary outcome of this study), as measured by the Functional Assessment Measure (FAM), compared to a control group receiving a standard paper-based program.

DETAILED DESCRIPTION:
All patients admitted to the NRZ receive a Baseline Assessment (T0). Rehabilitation aims are defined based on symptoms, functional limitations and participation restrictions, and routine care is provided accordingly. At discharge, patients undergo another assessment to determine if the rehabilitation aims have been reached (Post-inpatient Evaluation [T1]). Between T0 and T1, patients participating in this study will be randomly assigned to either a tele-reha group (Intervention Group) or a control group (Control Group 1) stratified for the likelihood of a positive rehabilitation outcome (determined by the multidisciplinary team), as well as age, and sex. Participation in the tele-reha group and the control group 1 is restricted to patients with SVS insurance. Additionally, a second control group (Control Group 2) will be recruited from patients without SVS insurance who only receive standard care. Control group 2 will be matched with the tele-reha group in terms of age group, sex and the likelihood of a positive rehabilitation outcome as estimated by the multidisciplinary team.

The study concludes with a final assessment (Final Evaluation) after 36 days of therapy. SVS patients from control group 1 will be offered the opportunity to participate in an additional tele-care intervention after the study ends. "EvoCare" is the platform for implementing the tele-care intervention, with most of the therapeutic content, such as exercise and training videos, produced by the NRZ. In addition, therapeutic content with a focus on cognition is entered into EvoCare and made available. Interventions will be selected based on the patient's primary concern in therapy, with a maximum of two activity goals and a maximum of two treatment foci set. Patients assigned to one of the control groups will continue with the standard care procedure, consisting of a paper-based home-exercise programme provided by the NRZ after discharge from the rehabilitation centre. This intervention is a programme of exercises for the basic motor skills of mobility, sensitivity, strength, endurance, balance and coordination. The supervising therapists select the content during the inpatient treatment and relate it to the patient's structural and activity-related limitations. The patients are given this paper-based programme at the end of their stay and then perform the exercises independently at home without further support.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older,
* experiencing problems with motor function, sensory function, cognition, swallowing or speech production (regardless of their diagnosis),
* being insured with SVS,
* agreeing to telerehabilitation after discharge,
* having sufficient motor and cognitive abilities to operate a smartphone, tablet or PC, or being sufficiently supported by caregivers, and
* being able to independently perform the targeted tasks assigned to them.

Exclusion Criteria:

- pronounced impairments in awareness, memory, attention, spatial performance, executive performance, apraxia, speech, and visual perception that do not allow a safe study participation according to the treating physicians or therapists

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in the Functional Assessment Measure (Changes from baseline measurement to evaluation at the end of inpatient rehabilitation to evaluation after the tele-rehab intervention) | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1), Evaluation after tele-reha up to 10 weeks after T1 (T2)
  Score 18-126 (higher score indication better functioning in everyday life)

SECONDARY OUTCOMES:
Quality of Life Measure | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  Numeric Rating Scale (NRS) 0-100 (higher score indicating better quality of life)
Pain level at the moment | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  NRS 0-100 (higher score indicating more symptomatology)
Pain level on average in the last weeks | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  NRS 0-100 (higher score indicating more symptomatology)
Health Status | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  NRS 0-100 (higher score indicating better health status)
Center for Epidemiologic Studies Depression Scale (CESD) | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  0-60 (higher socre indicating more symptomatology)
ZUF 8 Patient satisfaction | Baseline evaluation at start of inpatient rehabilitation (in protocol referred to as T0), Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1) , Evaluation after tele-reha up to 10 weeks after T1 (T2)
  1-4 (score varies according to questions)
Goal achievement scale | Evaluation at the end of inpatient rehabilitation up to 12 Weeks after T0 (in protocol referred to as T1), Evaluation after tele-reha up to 10 weeks after T1 (T2)
  1-5 (higher score indicating worse goal achievement)
Experience with tele-care | Evaluation after tele-reha up to 10 weeks after T1 (in protocol referred to asT2)
  1-4 (score varies according to questions)
Experience with standard care | Evaluation after tele-reha up to 10 weeks after T1 (in protocol referred to as T2)
  1-4 (score varies according to questions)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No